CLINICAL TRIAL: NCT05723770
Title: Effects of NOV03 on the Tear Film in Subjects With Dry Eye Disease
Brief Title: Effects of NOV03 on the Tear Film
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 922
Record Dates: First submitted 2023-01-19; First posted 2023-02-13 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: This pilot, open label, single-arm, single-center study will consist of 2 study visits in subjects with dry eye disease associated with MGD. A Screening Visit will occur to verify subjects are eligible to participate followed by an Assessment Visit to evaluate tear film parameters at baseline and over approx. 4 hours following a single instillation of NOV03
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Perfluorohexyloctane (Experimental)
  Interventions: Drug: instillation of NOV03

INTERVENTIONS:
Drug: instillation of NOV03 — This trial consists of 2 office visits over a period of approximately 2 weeks. At Visit 2, a designated clinical staff member or the investigator will instill 1 drop of NOV03 into each eye.

SUMMARY:
Determine the effect of a single instillation of NOV03 on the thickness and evaporation rate of the mucus-aqueous layer of the tear film

ELIGIBILITY:
Inclusion Criteria:

General/Ocular Inclusion Criteria

1. Will be at least 18 years of age at the time of consent. 2. Able to provide written voluntary informed consent. 3. Have a subject-reported history of DED in both eyes for at least 6 months prior to Visit 1. 4. Have Tear film break-up time (TFBUT) ≤5 sec at Visit

* Have Ocular Surface Disease Index (OSDI) ≥25 at Visit 1.
* Have an unanesthetized Schirmer's Test I ≥5 mm at Visit 1.
* Have Meibomian Gland Dysfunction (MGD) defined as total MGD score ≥ 3 (secretion of 5 central glands on lower eyelid will be evaluated, each will be scored from 0-3; 0 = normal, 1 = thick/yellow, whitish, particulate 2 = paste; 3 = none/occluded; total score will range from 0-15) at Visit 1.
* Have a total corneal fluorescein staining score of ≥2 and ≤11 (i.e. sum of inferior, superior, central, nasal, and temporal) according to the National Eye Institute (NEI) scale at Visit 1.
* Have at least one eye that satisfies all criteria for 4-8 above at Visit 1.
* Is able to fix his/her gaze for a minute, i.e. can see the fixation target and with no nystagmus
* Is able and willing to follow instructions, including participation in all trial assessments and visits.

Exclusion Criteria:

General/Ocular Exclusion Criteria

1. Have any clinically significant ocular surface slit-lamp findings at Visit 1 and Visit 2 and/or in the opinion of the Investigator had any findings that may have interfered with trial parameters, including

   1. history of eye trauma
   2. history of Stevens-Johnson syndrome
   3. active blepharitis or lid margin inflammation
   4. DED secondary to scarring, irradiation, alkali burns, cicatricial pemphigoid, or destruction of conjunctival goblet cells (as with vitamin A deficiency).
   5. abnormal lid anatomy that caused incomplete eyelid closure
   6. abnormal cornea shape (keratoconus)
   7. corneal epithelial defect or significant confluent staining or filaments
   8. history of herpetic keratitis.
   9. has a pterygium in either eye.
   10. ocular or periocular rosacea that in the judgement of the Investigator interfered with the trial
2. Has used any topical ocular steroids treatments, prescription dry eye therapy including varenicline nasal spray, or topical anti-glaucoma medication within 60 days prior to Visit 1.
3. Have had a LipiFlow procedure, intense pulse light procedure or any kind of other procedure affecting meibomian glands within 6 months prior to Visit 2.
4. Have received or removed a permanent punctum plug within 3 months (6 months for dissolvable punctum plugs) prior to Visit 2.
5. Have used any eye drops (prescription or artificial tears) and/or TrueTearTM device (intranasal tear neurostimulator) within 24 hours before Visit 2.
6. Have active ocular allergies or ocular allergies that are expected to be active during the trial period.
7. Have worn contact lenses within 1 month of Visit 1 or anticipate using contact lenses during the trial.
8. Have undergone intraocular surgery or ocular laser surgery within the previous 6 months or had any planned ocular and/or lid surgeries over the trial period.
9. Have an active ocular or systemic infection (bacterial, viral, or fungal), including fever requiring treatment with antibiotics.
10. Is a woman who was pregnant, nursing or planning a pregnancy.
11. Is a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception included: hormonal (oral, implantable, injectable, or transdermal contraceptives); mechanical (spermicide in conjunction with a barrier such as a diaphragm or condom); intrauterine device; or surgical sterilization of partner. For non-sexually active females, abstinence could have been regarded as an adequate method of birth control; however, if the subject becomes sexually active during the trial, she must agree to use adequate birth control as defined above for the remainder of the trial.
12. Has an uncontrolled systemic disease in the opinion of the Investigator will interfere with the trial.
13. Has a known allergy and/or sensitivity to the investigational drug.
14. Has used any oral medications known to cause ocular drying (e.g., antihistamines, antidepressants, etc.) on a non-stable regimen within 1 month prior to Visit 1 or is expected to be unstable during the trial.
15. Have taken isotretinoin (e.g. Accutane, Myorisan, Claravis, Amnesteem) within 6 months of Visit 1.
16. Has corrected VA worse than or equal to logarithm of the minimum angle of resolution (LogMAR), +0.7 as assessed with Early Treatment Diabetic Retinopathy Study (ETDRS) charts in both eyes at Visit 1.
17. Is currently enrolled in an investigational drug or device study or had used an investigational drug or device within 60 days of Visit 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 101, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Perfluorohexyloctane
Started | 33
Completed | 27
Not Completed | 6
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Perfluorohexyloctane
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 11
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Thickness of the Mucus-aqueous Tear Film Layer
Description: Thickness of the mucus-aqueous layer of the tear film, measured in nanometers
Time Frame: over 4 hours following instillation of NOV03
Population: The study had substantial technical data collection issues that prevented many of the subjects' parameter scores from being saved and analyzed. For the mucus-aqueous layer thickness the number of study eyes for which measurements were collected ranged from 15-24 rather than the planned 30 study eyes. Analysis was conducted without imputation of data. Thus, results were inconclusive due to data collection issues.
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Perfluorohexyloctane
Number analyzed (Participants) | 27
nm | 3920.3 (797.7)

2. Primary Outcome: Thinning Rate of the Mucus-aqueous Tear Film Layer
Description: The rate of change in the thickness of the tear film mucus-aqueous layer, measured in nanometers/second
Time Frame: over 4 hours following instillation of NOV03
Population: The study had substantial technical data collection issues that prevented many of the subjects' parameter scores from being saved and analyzed. For the mucus-aqueous layer thickness thinning rate (MALTR) the number of study eyes for which measurements were collected ranged from 6-11 rather than the planned 30 study eyes. Analysis was conducted without imputation of data. Thus, results were inconclusive due to data collection issues.
Measure: Mean (Standard Deviation); unit: nm/s
Arm/Group | Perfluorohexyloctane
Number analyzed (Participants) | 27
nm/s | -62.3 (90.9)

ADVERSE EVENTS:
Time Frame: Assessed for the entire study; Visit 1 Screening through Visit 2, an average of 2 weeks
Arm/Group | Perfluorohexyloctane
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

LIMITATIONS AND CAVEATS:
The study had substantial technical data collection issues that prevented many of the subjects' parameter scores from being saved and analyzed. In particular for the mucus-aqueous layer thickness thinning rate (MALTR) the number of study eyes for which measurements were collected ranged from 6-11 rather than the planned 30 study eyes. Analysis was conducted without imputation of data.Thus, results were inconclusive due to data collection issues and any representation of data would be misleading.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT05723770/Prot_SAP_002.pdf